CLINICAL TRIAL: NCT05946759
Title: Reoperation Rate in Breast-Conserving Surgery Using Confocal Histolog® Scanner for Intraoperative Margin Assessment in a Single-centric PMPF Study (SHIELD)
Brief Title: Reoperation Rate in Breast-Conserving Surgery Using Confocal Histolog® Scanner for Intraoperative Margin Assessment
Acronym: SHIELD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: SamanTree Medical SA (Industry)
Collaborators: St. Vincenz Krankenhaus GmbH, Paderborn (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: SHIELD
Record Dates: First submitted 2023-06-27; First posted 2023-07-14 (Actual); Last update posted 2024-03-21 (Actual); Status verified 2024-03

CONDITIONS: Breast Cancer - Ductal Carcinoma in Situ (DCIS); Breast-Conserving Surgery
Keywords: Reoperation Rate; Breast Conserving Surgery; Confocal laser scanning microscope; Confocal microscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Prospective (Active Comparator): 50 prospective subjects
  Interventions: Device: Histolog Scanner
- Historical (No Intervention): 40 historical subjects

INTERVENTIONS:
Device: Histolog Scanner — The PMPF study is collecting data that includes the use of the CE Mark IVD Histolog Scanner for the breast lumpectomy margin assessment.
  Arms: Prospective

SUMMARY:
This PMPF study is proposed to evaluate in real life the reoperation rates (ROR) of breast cancer and/or DCIS surgery when including the use of the HLS in the context of breast lumpectomy margin assessment.

ELIGIBILITY:
Inclusion Criteria:

* Adult female Subject ≥18 years old.
* Subject Scheduled for breast conserving surgery of invasive and/or in-situ ductal carcinoma.
* Subject is able to read, understand and sign the informed consent.

Exclusion Criteria:

* Subject previously treated for ipsilateral breast cancer and/or ductal carcinoma in situ surgery.
* Subject with previous radiotherapy of the ipsilateral breast.
* Subject with multicentric/multilateral breast cancer.
* Subject with planned mastectomy, tumor-adapted breast reduction.
* Subject with pre-surgical/ preoperative neo-adjuvant treatment.
* Subject is pregnant/ lactating.
* Participation in any other clinical study that would affect data acquisition.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2023-10-10 (Actual); Primary Completion 2024-03-12 (Actual); Study Completion 2024-03-12 (Actual)

PRIMARY OUTCOMES:
Reoperation Rate | 2-30 days post Breast Surgery
  Differences in the rate of reoperation due to cancer positive margins

SECONDARY OUTCOMES:
Margin status of intraoperative specimen vs. postoperative pathology assessment [Clinical Performance] | 0-30 days post Breast Surgery
  To observe real life clinical performance of the HLS and accessories when used intraoperatively
System Usability Scale (SUS) of the IVD device and accessories [Usability] | Only during the time of the breast surgery
  To survey usability of the HLS and accessories when used intraoperatively
Change in hospital cost with or without IVD device and accessories [Economic Impact] | 30 days post surgery date
  To evaluate the economic impact for the hospital/payer of the reoperation rate
Incidence of adverse device effects [Safety] | Only during the time of the breast surgery
  Incidence of adverse device effects during surgery

CONTACTS AND LOCATIONS:
Overall Officials: Michael P Lux, Prof. Dr MBA, Principal Investigator — St. Vincenz Krankenhaus GmbH, Paderborn
Locations (1):
- St. Vincenz-Krankenhaus GmbH, Frauenklinik St. Louise, Paderborn, Germany

IPD SHARING:
Plan to Share IPD: No